CLINICAL TRIAL: NCT06897280
Title: A Single-Center, Prospective Clinical Trial of MED HF10™ Spinal Cord Stimulation for the Treatment of Chronic Pain
Brief Title: Clinical Trial of MED HF10™ Spinal Cord Stimulation for the Treatment of Chronic Pain
Acronym: MED
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nevro Corp (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1309273; MED IIS (Other: Nevro Corp)
Record Dates: First submitted 2025-03-10; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Chronic, Intractable Back Pain And/or Leg Pain
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single arm (Experimental): Pulse Dosing
  Interventions: Device: SCS Device Program Setting

INTERVENTIONS:
Device: SCS Device Program Setting — A Pulse Dose setting specifies a brief duration of stimulation 'on' and stimulation 'off' durations, applied in a continuously cycled manner
  Other Names: Pulse Dose Setting

SUMMARY:
This is a single-center, prospective, non-randomized exploratory study in subjects with chronic, intractable back pain and/or leg pain per the center's routine practice. The primary endpoint is the distribution of responders by 'lowest preferred pulse dose (PD)' setting, where a subject is a responder to the lowest PD setting they preferred prior to entering the Observational period. The study is performed in patients who already have Nevro SCS devices implanted.

ELIGIBILITY:
Inclusion Criteria:

1. Have been diagnosed with chronic, intractable pain of the back pain with or without leg pain
2. Have been implanted with the Nevro Senza™ or Omnia SCS system with dual leads, approximately over vertebral T8-T11, for at least 3 months, and are using the system with single area, continuous 10 kHz stimulation programs at least 18 hours daily, as determined by subject reporting and confirmation via device diagnostics, for at least 21 days prior to enrolling in this study
3. If taking them, be on stable chronic pain medications, as determined by the Investigator, for at least 28 days prior to enrolling in the study and be willing to stay on those medications with no dose adjustments until study completion or study withdrawal, whichever comes first.
4. Be 18 years of age or older at the time of enrollment
5. Be willing and able to comply with study-related requirements, procedures, and visits
6. Be capable of subjective evaluation, able to read and understand IRB approved written questionnaires, and are able to read, understand and sign the IRB approved written informed consent, all of which will be in American English
7. Be compliant in using the patient programmer and recharger as determined by the Investigator.
8. As determined by the Investigator, be compliant in adjusting programs using the device remote control.
9. Have >= 30% pain relief in primary pain area intended to be treated by SCS.

Exclusion Criteria:

1. Have a medical condition or pain in other area(s), not intended to be treated with SCS, that could interfere with study procedures, accurate pain reporting, and/or confound evaluation of study endpoints, as
2. Have evidence of an active disruptive psychological or psychiatric disorder or other known condition significant enough to impact perception of pain, compliance of intervention and/or ability to evaluate treatment outcome.
3. Have a current diagnosis of a progressive neurological disease such as multiple sclerosis, chronic inflammatory demyelinating polyneuropathy, rapidly progressive arachnoiditis, rapidly progressive diabetic peripheral neuropathy, brain or spinal cord tumor, central deafferentation syndrome, Complex Regional Pain Syndrome, or acute herniating disc, as determined by the investigator.
4. Having any clinical evidence mechanical instability or progressive neurologic pathology that warrants surgical intervention.
5. Having undergone an interventional procedure and/or surgery to treat back or leg pain other than Senza HF10 therapy in the last 30 days
6. Have a condition currently requiring or likely to require diathermy
7. Have a condition currently requiring or likely to require surgery during the study period.
8. Have metastatic malignant disease or active local malignant disease
9. Have a life expectancy of less than 1 year
10. Have an active systemic or local infection
11. Be pregnant or planning to become pregnant during the course of the study (if female and sexually active, subject must be using a reliable form of birth control, be surgically sterile or be at least 2 years post-menopausal)
12. Have within 6 months of enrollment a significant untreated addiction to dependency producing medications or have been a substance abuser (including alcohol and illicit drugs)
13. Be concomitantly participating or planned to be participating in another clinical study overlapping in time with the present clinical study
14. Have an existing drug pump and/or another active implantable device (switched On or Off) such as a pacemaker or other non-Senza™ SCS devices
15. Have an unresolved condition of device-related pain (e.g. IPG pocket
16. Have a condition currently requiring or likely to require surgery during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2024-11-16 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Preference for Pulse Dose Setting | 3 months
  Starting from a standardized low pulse dose (PD) setting, subjects will try progressively lower PD settings depending upon their response to each setting, to arrive at the lowest PD setting they prefer. Up to 5 PD settings will be tried by each subject.

SECONDARY OUTCOMES:
Numerical Rating Scale of Back, Leg, and Overall Pain Intensity | 3 months
  The numerical rating scale ranges from 0 to 10, where 0 = no pain and 10 = worst pain imaginable.
Patient Satisfaction | 3 months
  The subject will rate their satisfaction with the SCS program on a scale from "Very Satisfied," "Satisfied," "Not Sure," "Dissatisfied," to "Very Dissatisfied."
Patient Global Impression of Change | 3 months
  This 7-point scale is used to assess the subject's global change in their general state of health for each particular phase of the study. Responses range from "Very Much Worse" to "No Change" to "A Great Deal Better".
Oswestry Disability Index | 3 months
  The Oswestry Disability Index (ODI) uses 10 questions covering aspects of daily life affected by back pain, such as pain intensity, personal care, lifting, walking, and social activities. Each question is scored on a 0-5 scale, with higher scores indicating greater disability. The total score is calculated as a percentage, with 0% representing no disability and 100% representing complete disability. Outcomes will be categorized as follows: 0-20%: Minimal disability; 21-40%: Moderate disability; 41-60%: Severe disability; 61-80%: Crippled; 81-100%: Bedridden.
Patient Catastrophizing Scale | 3 months
  Subjects are asked to indicate the degree to which they have the above thoughts and feelings when they are experiencing pain using the 0 (not at all) to 4 (all the time) scale. A total score is yielded (ranging from 0-52), along with three subscale scores assessing rumination, magnification and helplessness.
PROMIS-SF Sleep Disturbance Scale | 3 months
  Each of the 8 items on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 8 to 40 with higher scores indicating greater severity of sleep disturbance.
Daily device recharge duration | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mayank Gupta, MD, Principal Investigator — Neuroscience Research Center
Locations (1):
- Neuroscience Research Center, Overland Park, Kansas, United States